CLINICAL TRIAL: NCT02260128
Title: Effect of Chewing Gum on Postoperative Bowel Function Following Upper GI Tract Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Michael Bau Mortensen (Other)
Responsible Party: Sponsor-Investigator, Michael Bau Mortensen, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tyggegummi
Record Dates: First submitted 2014-10-05; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Cancer Esophagus; Pancreatic Cancer
Keywords: postoperative ileus; chewing gum
MeSH Terms: conditions — Esophageal Neoplasms; Pancreatic Neoplasms | interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gum chewing (Experimental): This intervention group will receive chewing gum four times daily following surgery. Each of which they are encouraged to chew for 30 minutes.
  Gum chewing is terminated when one of the primary end points occurs.
  Interventions: Other: Chewing gum
- Control group (No Intervention): This group will receive the normal postoperative treatment. Occurence of primary end points are registrered.

INTERVENTIONS:
Other: Chewing gum — The intervention group will receive chewing gum four times daily following surgery.
  Arms: Gum chewing

SUMMARY:
Every patient undergoing surgery in the abdomen will experience temporary paralysis of bowel function. This study evaluates whether chewing gum can reduce the bowel paralysis after surgery in patients undergoing either esophageal resection or whipples procedure. Half the study population will receive chewing gum while the other half will act as control.

DETAILED DESCRIPTION:
Every surgical procedure results in a temporary paralysis of bowel function. This condition is named postoperative ileus (POI) and it is characterized by absence of intestine motility, accumulation of gas and fluid inside the intestines and absence of flatus and defecation. It results in nausea, vomiting, abdominal distension, pain and lowered tolerance towards intake of fluid and solid foods. POI is the organism's reaction to the surgical trauma and it is most often the single most important factor determining the length of patient admission. Prolonged POI can also result in medical complications.

The length of POI following elective abdominal surgery is most often 3 to 6 days. Gradually during this period the intestines regain their normal behavioral pattern. The colon is the last segment to regain its motility which decides the patient's wellbeing. Therefore most investigations of POI measure time from surgery to first flatus or defecation.

The cause of POI is found in the surgical trauma. When the abdominal wall and the peritoneum are penetrated and the intestines exposed and handled, the immune system is activated. The immune system creates an inflammatory response that inhibits the local neural pathways in the intestines. The size of the immune response is related to the size of the surgical procedure and the length of POI. Together with the overall hormonal surgical stress response the inflammatory response creates a shift in the autonomous nervous system towards sympathetic domination. This further inhibits bowel activity.

The intake of food activates parasympathetic activity and promotes bowel activity. Early food intake following abdominal surgery, however, is often ill received by the patients hence the above mentioned symptoms of POI. The early food intake can also worsen complications following surgery such as anastomotic leakage. This is most pronounced with anastomoses on the esophagus and stomach. Therefore abstinence from food intake is often recommended in the immediate postoperative period.

Chewing of chewing gum following surgery can be perceived as placebo intake of food because it also activates the parasympathetic nervous system and under normal conditions the cephalic part of the digestion. Gum chewing does not, however, result in worsening of potential surgical complications and it is generally well tolerated by the patients. Postoperative gum chewing has been investigated and found effect full in the shape of reduced POI following colorectal surgery, abdominal surgery on the aorta, bladder surgery, and caesarian section.

The effect of gum chewing following surgery on the esophagus and the pancreas has to our knowledge not yet been investigated.

With this study we wish to investigate the effect of gum chewing on POI in a patient population undergoing either esophageal resection or pancreaticoduodenectomy (whipples procedure) due to cancer in either the esophagus or the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing esophageal/cardial resection due to cancer and patients undergoing whipples procedure due to cancer.
* Macroradical resection must be accomplished.
* Informed consent given.

Exclusion Criteria:

* Patients WHO fail to follow the study regimen for more than 24 hours.
* Patients under the age of 18 years.
* Pregnant or beast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Time from surgery to first flatus | 7 days
Time from surgery to first defecation | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bau Mortensen, Professor, Principal Investigator — Departement of Surgery, Odense University Hospital
Locations (1):
- Department of Surgery, Odense University Hospital, Odense, Denmark